CLINICAL TRIAL: NCT03957265
Title: Prospective Observational Study of SynCone® Concept: Patient-related Outcomes, Clinical, Radiographic, Immunoinflammatory Mediators and Microbiological Analysis
Brief Title: Prospective Observational Study of SynCone® Concept
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marcio Zaffalon Casati (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor-Investigator, Marcio Zaffalon Casati, professor, Paulista University
Organization: Paulista University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79380717.4.0000.5512
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Jaw, Edentulous
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Syncone (Experimental): Tapered abutment connection
  Interventions: Procedure: Tapered abutment connection

INTERVENTIONS:
Procedure: Tapered abutment connection — Rehabilitation of completely edentulous patients with overdentures prostheses.

SUMMARY:
The aim of this prospective observational study will be to evaluate patient-related outcomes, clinical, microbiological and peri-implant immunoinflammatory mediators in completely edentulous patients rehabilitated with delayed loaded overdentures prostheses. The investigators hypothetize that this system could restore edentulous patients with healthier mucosal concerning clinical, microbiological and immunoinflammatory parameters, besides to promote improvement in patient satisfaction and quality of life.

DETAILED DESCRIPTION:
This prospective observational study will include fifteen edentulous patients rehabilitated with conventional dentures. Patients will receive four to six maxillary implants loaded three months after surgery. Clinical, microbiological and immunoinflammatory parameters will be evaluated at baseline, three, and six months following overdenture prosthesis. Patient-centered/reported outcomes concerning general satisfaction with the prostheses as well as comfort, ability to speak, stability, esthetics, ease of cleaning and occlusion, will be evaluated at baseline (conventional denture evaluation) and after 6 months (overdenture evaluation).

ELIGIBILITY:
Inclusion Criteria:

* subject has total edentulous maxilla.
* subject whose dental extractions occurred at least 6 months before treatment.

Exclusion Criteria:

* pregnancy, lactation, smoking or ex-smokers, systemic conditions that could affect bone metabolism (e.g., immunologic disorders, diabetes), use of anti-inflammatory, biphosphonate, and immunosuppressive medications, subjects that required bone grafts before/during implant surgery.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2021-09-17 (Estimated); Study Completion 2022-03-17 (Estimated)

PRIMARY OUTCOMES:
Modified Gingival Index | 6 months
  Index of mucosal condition (Mombelli et al.1987): 0 - No bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant, 1 - Isolated bleeding spots visible, 2 - Blood forms a confluent red line on mucosal margin, 3 - Heavy or profuse bleeding

SECONDARY OUTCOMES:
Modified Plaque Index | 6 months
  Index of plaque accumulation (Mombelli et al.1987): 0 - No detection of plaque, Plaque only recognized by running a probe accross the smooth marginal surface of the implant, 2 - Plaque can be seen by the naked eye, 3 - Abundance of soft matter.
Oral Healthy Impact Profile-14 (OHIP-14) | 6 months
  A questionnaire will be administered to evaluate patient centered outcomes with regards to prosthesis. It has 14 questions in which the patient answers between never (0), rarely (1), sometimes (2), repeatedly (3) and always (4).
Microbiological assays | 6 months
  Peri-implant biofilm will be collected and Real Time PCR wil be performed to measure the absolute quantification of Aggregatibacter Actinomycetemcomitans, Porphyromonas gingivalis, and Tannerella forsythensis
Concentration of osteoimmuneinflammatory mediators | 6 months
  Levels of osteoimmuneinflammatory mediators will be determined in the peri-implant fluid (IL-4, IL-17, IL-1β, IL-10, IL-6, IL-8, IL-23 and TNF-α)
Crestal bone level | 6 months
  Periapical radiographs will be made to evaluate crestal bone level alteration.

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry - Paulista University UNIP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No